CLINICAL TRIAL: NCT06668922
Title: Fecal Bile Acids, Fecal Short Chain Fatty Acids and the Intestinal Microbiota in Patients With Irritable Bowel Syndrome (IBS) and Control Volunteers: Diet Challenge
Brief Title: Irritable Bowel Syndrome and Control Volunteers: Diet Challenge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrea S. Shin, MD, Associate Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-0442
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: irritable bowel syndrome; IBS; short-chain fatty acids; SCFAs; bile acids; fecal inulin; microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Experimental): Adults ages 18-65 years with no prior history of gastrointestinal diseases or symptoms.
  Interventions: Dietary Supplement: Inulin
- Irritable Bowel Syndrome Patients with Diarrhea (IBS-D) (Experimental): Patients with irritable bowel syndrome (IBS) with diarrhea, ages 18-65 years fulfilling Rome IV criteria for IBS.
  Interventions: Dietary Supplement: Inulin
- Irritable Bowel Syndrome Patients with Constipation (IBS-C) (Experimental): Patients with irritable bowel syndrome (IBS) with constipation, ages 18-65 years fulfilling Rome IV criteria for IBS.
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Inulin ingestion is not being used to diagnose, treat, or prevent IBS. Inulin is being used to study an individual's ability to ferment dietary fiber.

SUMMARY:
The study will investigate the relationship between fecal bile acids, short-chain fatty acids (SCFAs), and the gut microbiota in irritable bowel syndrome (IBS). The central hypothesis of this study is that specific shifts in the GI microbiome composition correlate with altered colonic SCFAs and BAs and contribute to IBS symptoms. Primary aims include: (a) identifying GI microbiome signatures in IBS subtypes (IBS-C and IBS-D) and matched controls, and test if microbiome signatures in these groups correlate with fecal SCFAs and bacterial fermentation of an indigestible carbohydrate (inulin) after a dietary challenge (fecal inulin), and (b) determining if GI microbiome signatures in IBS subtypes and controls correlate with fecal BAs or markers of SCFA production (fecal SCFAs or inulin) and test if BAs correlate with fecal SCFAs or inulin.

The target population is adults ages 18-65 years meeting Rome IV criteria for IBS (both diarrhea- and constipation-predominant, IBS-D and IBS-C) and asymptomatic controls. Primary outcomes will be fecal bile acid excretion and profile, short-chain fatty acid excretion and profile, colonic transit, and fecal microbiota. Secondary outcomes will be stool characteristics based on responses to validated bowel diaries. Stool samples will be collected from participants during the last 2 days of a 4-day 100 g fat diet and split into 3 samples for fecal microbiota, SCFA, and bile acid analysis.

DETAILED DESCRIPTION:
During the study:

Screening/Visit 1

* Participants will be asked to read and sign this informed consent after all questions about the study have been answered to satisfaction.
* This is a screening visit, and we may determine that a participant is ineligible to continue to participate in the study.
* The study team will collect medication and medical history.
* A physical exam will be performed by the physician. Vital signs and body measurements will be collected.
* Participants will be provided with a take-home lasagna meal (vegetarian and non-vegetarian option) and dessert.
* Participants will receive a stool collection kit and instructions for the collection, storage, and transportation of stool.
* Instructions will be provided for a low fiber, high fat diet for Days 2-4.
* Participants will be asked to complete diet recall using the ASA24 and a bowel pattern diary to record bowel symptoms over the course of the study.
* IBS participants will complete the irritable bowel syndrome severity scoring system questionnaires (IBS-SSS).

Day 2-4 (at home):

* Participants will record stool symptoms and patterns in a diary daily.
* Participants will be instructed to consume a low fiber diet (maximum one piece of fruit and 100 g of vegetables a day, and white flour instead of whole grain products), avoid alcohol, and start a 4-day 100 g fat diet.
* On the evening before Day 5, participants will be instructed to collect a stool sample at home and return during Visit 2.

Day 5 (Visit 2):

* Participants will return to the clinic on Day 5 after an overnight fast.
* Participants in the reproductive age range will be given a urine pregnancy test prior to inulin ingestion and the study team will confirm a negative test result.
* Participants will receive breakfast onsite. The non-vegetarian option will consist of pancakes, butter, syrup, hard-boiled eggs, and bacon. The vegetarian option will substitute the bacon with a cheese snack (approximately 790 to 840 kcal) along with 10 g inulin Orafti® powder) thoroughly mixed in 200 mL of water.
* Take-home meals will be provided for lunch and dinner and are to be consumed at 4 and 8 hours from breakfast.
* IBS participants will complete the irritable bowel syndrome severity scoring system (IBS-SSS) questionnaire.
* A stool sample will be collected on Day 5.
* Participants will continue to complete diet recall using the ASA24 and a bowel pattern diary to record bowel symptoms over the course of the study.

Day 6

* Participants will be instructed to collected a final stool sample (Day 6).
* Participants will continue to complete diet recall using the ASA24 and a bowel pattern diary to record bowel symptoms over the course of the study.

Day 7 (Visit 3)

• Participants will return to the clinic to return stool collections (Day 5 and Day 6), the daily diaries, and the IBS-SSS forms (if applicable).

Day 30-90 (Optional dietary follow-up): To further assess the utility of the 24 hour dietary recall, willing participants will be invited to participate in a an optional follow-up activity during which they will complete the Automated Self-Administered Dietary Assessment Tool with or without assistance of a trained interviewer. Interested volunteers will be contacted by phone and provided instructions on how to complete the tool online by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Individuals with irritable bowel syndrome (IBS)
* Healthy volunteers (healthy controls) with no prior history of gastrointestinal (GI) disease or symptoms
* No dietary restrictions other than vegetarian

Exclusion Criteria:

* Inflammatory bowel disease, celiac disease, or certain types of abdominal cancer, as well as those with thyroid or liver issues
* Abdominal surgery or abdominal radiation within 6 months of study participation, with an exception for C-section or gallbladder removal
* Use of any prescription, over the counter, or herbal medications known to affect gastrointestinal function or study interpretation, such as opioids, inflammatory drugs or certain antidepressants, within 6 months prior to study participation for healthy volunteers, or within 2 days of study participation for participants with IBS.
* An exception will be permitted for limited use of stable low doses of antidepressants for individuals who have been taking them for a period greater than one month.
* Rescue medication such as Bisacodyl (dulcolax) to relieve severe constipation and allow for stool collection will be permitted when needed.
* Use of Ozempic and Ozempic-type medications
* Pregnant or breastfeeding women
* Antibiotic use within 3 months of study participation
* Use of prebiotics or probiotics within the 2 weeks before the study initiation
* Regular tobacco use within the past 6 months

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Total fecal bile acids | 48 hours
  Stool samples will be collected over 2 days for measurement of fecal bile acids (µmol/48h) by high performance liquid chromatography-mass spectometry.
Total fecal short chain fatty acids | 48 hours
  Stool samples will be collected for measurement of measurement of short chain fatty acids (µg/mg) by liquid chromatography-mass spectrometry
Individual fecal short chain fatty acids | 48 hours
  Stool samples will be collected for measurement of measurement of short chain fatty acids (µg/mg) by liquid chromatography-mass spectrometry
Fecal microbial population | 48 hours
  Stool samples will be be collected from participants for nucleic acid extraction, 16S allele PCR and sequencing to measure microbial communities and profiles of specimens
Fecal inulin | 48 hours
  Fecal inulin content will be measured using short acid hydrolysis and high-performance liquid chromatography

SECONDARY OUTCOMES:
Percent primary fecal bile acids | 48 hours
  Stool samples will be collected over 2 days for measurement of fecal bile acids (µmol/48h) by high performance liquid chromatography-mass spectrometry.
Stool characteristics | 4 days
  Stool characteristics will be measured using a 4 day bowel diary

OTHER OUTCOMES:
24-hour diet (food intake) recall | 6 days
  24-hour dietary intake will be submitted using web-based Automated Self-Administered Dietary Assessment Tool developed by the National Cancer Institute (https://epi.grants.cancer.gov/asa24/).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Wong BS, Camilleri M, McKinzie S, Burton D, Graffner H, Zinsmeister AR. Effects of A3309, an ileal bile acid transporter inhibitor, on colonic transit and symptoms in females with functional constipation. Am J Gastroenterol. 2011 Dec;106(12):2154-64. doi: 10.1038/ajg.2011.285. Epub 2011 Aug 30. PMID 21876564
- [Background] Chey WD, Camilleri M, Chang L, Rikner L, Graffner H. A randomized placebo-controlled phase IIb trial of a3309, a bile acid transporter inhibitor, for chronic idiopathic constipation. Am J Gastroenterol. 2011 Oct;106(10):1803-12. doi: 10.1038/ajg.2011.162. Epub 2011 May 24. PMID 21606974
- [Background] Walters JR, Johnston IM, Nolan JD, Vassie C, Pruzanski ME, Shapiro DA. The response of patients with bile acid diarrhoea to the farnesoid X receptor agonist obeticholic acid. Aliment Pharmacol Ther. 2015 Jan;41(1):54-64. doi: 10.1111/apt.12999. Epub 2014 Oct 20. PMID 25329562
- [Background] Musch MW, Bookstein C, Xie Y, Sellin JH, Chang EB. SCFA increase intestinal Na absorption by induction of NHE3 in rat colon and human intestinal C2/bbe cells. Am J Physiol Gastrointest Liver Physiol. 2001 Apr;280(4):G687-93. doi: 10.1152/ajpgi.2001.280.4.G687. PMID 11254495
- [Background] Murray RD, McClung HJ, Li BU, Ailabouni A. Stimulatory effects of short-chain fatty acids on colonic absorption in newborn piglets in vivo. J Pediatr Gastroenterol Nutr. 1989 Jan;8(1):95-101. doi: 10.1097/00005176-198901000-00018. PMID 2732869
- [Background] Fukumoto S, Tatewaki M, Yamada T, Fujimiya M, Mantyh C, Voss M, Eubanks S, Harris M, Pappas TN, Takahashi T. Short-chain fatty acids stimulate colonic transit via intraluminal 5-HT release in rats. Am J Physiol Regul Integr Comp Physiol. 2003 May;284(5):R1269-76. doi: 10.1152/ajpregu.00442.2002. PMID 12676748
- [Background] Mitsui R, Ono S, Karaki S, Kuwahara A. Neural and non-neural mediation of propionate-induced contractile responses in the rat distal colon. Neurogastroenterol Motil. 2005 Aug;17(4):585-94. doi: 10.1111/j.1365-2982.2005.00669.x. PMID 16078948
- [Background] Banasiewicz T, Krokowicz L, Stojcev Z, Kaczmarek BF, Kaczmarek E, Maik J, Marciniak R, Krokowicz P, Walkowiak J, Drews M. Microencapsulated sodium butyrate reduces the frequency of abdominal pain in patients with irritable bowel syndrome. Colorectal Dis. 2013 Feb;15(2):204-9. doi: 10.1111/j.1463-1318.2012.03152.x. PMID 22738315
- [Background] Mortensen PB, Andersen JR, Arffmann S, Krag E. Short-chain fatty acids and the irritable bowel syndrome: the effect of wheat bran. Scand J Gastroenterol. 1987 Mar;22(2):185-92. doi: 10.3109/00365528708991878. PMID 3033815
- [Background] Tana C, Umesaki Y, Imaoka A, Handa T, Kanazawa M, Fukudo S. Altered profiles of intestinal microbiota and organic acids may be the origin of symptoms in irritable bowel syndrome. Neurogastroenterol Motil. 2010 May;22(5):512-9, e114-5. doi: 10.1111/j.1365-2982.2009.01427.x. Epub 2009 Nov 10. PMID 19903265
- [Background] Treem WR, Ahsan N, Kastoff G, Hyams JS. Fecal short-chain fatty acids in patients with diarrhea-predominant irritable bowel syndrome: in vitro studies of carbohydrate fermentation. J Pediatr Gastroenterol Nutr. 1996 Oct;23(3):280-6. doi: 10.1097/00005176-199610000-00013. PMID 8890079
- [Background] Aguilera M, Cerda-Cuellar M, Martinez V. Antibiotic-induced dysbiosis alters host-bacterial interactions and leads to colonic sensory and motor changes in mice. Gut Microbes. 2015;6(1):10-23. doi: 10.4161/19490976.2014.990790. Epub 2015 Jan 20. PMID 25531553
- [Background] Jalanka-Tuovinen J, Salojarvi J, Salonen A, Immonen O, Garsed K, Kelly FM, Zaitoun A, Palva A, Spiller RC, de Vos WM. Faecal microbiota composition and host-microbe cross-talk following gastroenteritis and in postinfectious irritable bowel syndrome. Gut. 2014 Nov;63(11):1737-45. doi: 10.1136/gutjnl-2013-305994. Epub 2013 Dec 5. PMID 24310267
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Simren M, Brazier J, Coremans G, Dapoigny M, Muller-Lissner SA, Pace F, Smout AJ, Stockbrugger RW, Vatn MH, Whorwell PJ. Quality of life and illness costs in irritable bowel syndrome. Digestion. 2004;69(4):254-61. doi: 10.1159/000079846. Epub 2004 Jul 14. PMID 15256832
- [Background] Wedlake L, A'Hern R, Russell D, Thomas K, Walters JR, Andreyev HJ. Systematic review: the prevalence of idiopathic bile acid malabsorption as diagnosed by SeHCAT scanning in patients with diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2009 Oct;30(7):707-17. doi: 10.1111/j.1365-2036.2009.04081.x. Epub 2009 Jun 30. PMID 19570102
- [Background] Gracie DJ, Kane JS, Mumtaz S, Scarsbrook AF, Chowdhury FU, Ford AC. Prevalence of, and predictors of, bile acid malabsorption in outpatients with chronic diarrhea. Neurogastroenterol Motil. 2012 Nov;24(11):983-e538. doi: 10.1111/j.1365-2982.2012.01953.x. Epub 2012 Jul 5. PMID 22765392
- [Background] Shin A, Camilleri M, Vijayvargiya P, Busciglio I, Burton D, Ryks M, Rhoten D, Lueke A, Saenger A, Girtman A, Zinsmeister AR. Bowel functions, fecal unconjugated primary and secondary bile acids, and colonic transit in patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1270-1275.e1. doi: 10.1016/j.cgh.2013.04.020. Epub 2013 Apr 30. PMID 23639599
- [Background] Alemi F, Poole DP, Chiu J, Schoonjans K, Cattaruzza F, Grider JR, Bunnett NW, Corvera CU. The receptor TGR5 mediates the prokinetic actions of intestinal bile acids and is required for normal defecation in mice. Gastroenterology. 2013 Jan;144(1):145-54. doi: 10.1053/j.gastro.2012.09.055. Epub 2012 Oct 3. PMID 23041323
- [Background] Mroz MS, Keating N, Ward JB, Sarker R, Amu S, Aviello G, Donowitz M, Fallon PG, Keely SJ. Farnesoid X receptor agonists attenuate colonic epithelial secretory function and prevent experimental diarrhoea in vivo. Gut. 2014 May;63(5):808-17. doi: 10.1136/gutjnl-2013-305088. Epub 2013 Aug 5. PMID 23916961
- [Background] Marshall JK, Thabane M, Garg AX, Clark WF, Salvadori M, Collins SM; Walkerton Health Study Investigators. Incidence and epidemiology of irritable bowel syndrome after a large waterborne outbreak of bacterial dysentery. Gastroenterology. 2006 Aug;131(2):445-50; quiz 660. doi: 10.1053/j.gastro.2006.05.053. PMID 16890598
- [Background] Neal KR, Hebden J, Spiller R. Prevalence of gastrointestinal symptoms six months after bacterial gastroenteritis and risk factors for development of the irritable bowel syndrome: postal survey of patients. BMJ. 1997 Mar 15;314(7083):779-82. doi: 10.1136/bmj.314.7083.779. PMID 9080994
- [Background] Taverniti V, Guglielmetti S. Methodological issues in the study of intestinal microbiota in irritable bowel syndrome. World J Gastroenterol. 2014 Jul 21;20(27):8821-36. doi: 10.3748/wjg.v20.i27.8821. PMID 25083056
- [Background] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Background] Shukla R, Ghoshal U, Dhole TN, Ghoshal UC. Fecal Microbiota in Patients with Irritable Bowel Syndrome Compared with Healthy Controls Using Real-Time Polymerase Chain Reaction: An Evidence of Dysbiosis. Dig Dis Sci. 2015 Oct;60(10):2953-62. doi: 10.1007/s10620-015-3607-y. Epub 2015 Mar 18. PMID 25784074
- [Background] Lyra A, Rinttila T, Nikkila J, Krogius-Kurikka L, Kajander K, Malinen E, Matto J, Makela L, Palva A. Diarrhoea-predominant irritable bowel syndrome distinguishable by 16S rRNA gene phylotype quantification. World J Gastroenterol. 2009 Dec 21;15(47):5936-45. doi: 10.3748/wjg.15.5936. PMID 20014457
- [Background] Sundin J, Rangel I, Fuentes S, Heikamp-de Jong I, Hultgren-Hornquist E, de Vos WM, Brummer RJ. Altered faecal and mucosal microbial composition in post-infectious irritable bowel syndrome patients correlates with mucosal lymphocyte phenotypes and psychological distress. Aliment Pharmacol Ther. 2015 Feb;41(4):342-51. doi: 10.1111/apt.13055. Epub 2014 Dec 18. PMID 25521822
- [Background] Carroll IM, Ringel-Kulka T, Keku TO, Chang YH, Packey CD, Sartor RB, Ringel Y. Molecular analysis of the luminal- and mucosal-associated intestinal microbiota in diarrhea-predominant irritable bowel syndrome. Am J Physiol Gastrointest Liver Physiol. 2011 Nov;301(5):G799-807. doi: 10.1152/ajpgi.00154.2011. Epub 2011 Jul 7. PMID 21737778
- [Background] Pozuelo M, Panda S, Santiago A, Mendez S, Accarino A, Santos J, Guarner F, Azpiroz F, Manichanh C. Reduction of butyrate- and methane-producing microorganisms in patients with Irritable Bowel Syndrome. Sci Rep. 2015 Aug 4;5:12693. doi: 10.1038/srep12693. PMID 26239401
- [Background] Rajilic-Stojanovic M, Biagi E, Heilig HG, Kajander K, Kekkonen RA, Tims S, de Vos WM. Global and deep molecular analysis of microbiota signatures in fecal samples from patients with irritable bowel syndrome. Gastroenterology. 2011 Nov;141(5):1792-801. doi: 10.1053/j.gastro.2011.07.043. Epub 2011 Aug 5. PMID 21820992
- [Background] Rigsbee L, Agans R, Shankar V, Kenche H, Khamis HJ, Michail S, Paliy O. Quantitative profiling of gut microbiota of children with diarrhea-predominant irritable bowel syndrome. Am J Gastroenterol. 2012 Nov;107(11):1740-51. doi: 10.1038/ajg.2012.287. PMID 22986438
- [Background] Carroll IM, Ringel-Kulka T, Siddle JP, Klaenhammer TR, Ringel Y. Characterization of the fecal microbiota using high-throughput sequencing reveals a stable microbial community during storage. PLoS One. 2012;7(10):e46953. doi: 10.1371/journal.pone.0046953. Epub 2012 Oct 5. PMID 23071673
- [Background] Durban A, Abellan JJ, Jimenez-Hernandez N, Artacho A, Garrigues V, Ortiz V, Ponce J, Latorre A, Moya A. Instability of the faecal microbiota in diarrhoea-predominant irritable bowel syndrome. FEMS Microbiol Ecol. 2013 Dec;86(3):581-9. doi: 10.1111/1574-6941.12184. Epub 2013 Aug 23. PMID 23889283
- [Background] Carroll IM, Ringel-Kulka T, Siddle JP, Ringel Y. Alterations in composition and diversity of the intestinal microbiota in patients with diarrhea-predominant irritable bowel syndrome. Neurogastroenterol Motil. 2012 Jun;24(6):521-30, e248. doi: 10.1111/j.1365-2982.2012.01891.x. Epub 2012 Feb 20. PMID 22339879
- [Background] Malinen E, Krogius-Kurikka L, Lyra A, Nikkila J, Jaaskelainen A, Rinttila T, Vilpponen-Salmela T, von Wright AJ, Palva A. Association of symptoms with gastrointestinal microbiota in irritable bowel syndrome. World J Gastroenterol. 2010 Sep 28;16(36):4532-40. doi: 10.3748/wjg.v16.i36.4532. PMID 20857523
- [Background] Jeffery IB, O'Toole PW, Ohman L, Claesson MJ, Deane J, Quigley EM, Simren M. An irritable bowel syndrome subtype defined by species-specific alterations in faecal microbiota. Gut. 2012 Jul;61(7):997-1006. doi: 10.1136/gutjnl-2011-301501. Epub 2011 Dec 16. PMID 22180058
- [Background] Chassard C, Dapoigny M, Scott KP, Crouzet L, Del'homme C, Marquet P, Martin JC, Pickering G, Ardid D, Eschalier A, Dubray C, Flint HJ, Bernalier-Donadille A. Functional dysbiosis within the gut microbiota of patients with constipated-irritable bowel syndrome. Aliment Pharmacol Ther. 2012 Apr;35(7):828-38. doi: 10.1111/j.1365-2036.2012.05007.x. Epub 2012 Feb 8. PMID 22315951
- [Background] Duboc H, Rainteau D, Rajca S, Humbert L, Farabos D, Maubert M, Grondin V, Jouet P, Bouhassira D, Seksik P, Sokol H, Coffin B, Sabate JM. Increase in fecal primary bile acids and dysbiosis in patients with diarrhea-predominant irritable bowel syndrome. Neurogastroenterol Motil. 2012 Jun;24(6):513-20, e246-7. doi: 10.1111/j.1365-2982.2012.01893.x. Epub 2012 Feb 22. PMID 22356587
- [Background] Stephen AM, Haddad AC, Phillips SF. Passage of carbohydrate into the colon. Direct measurements in humans. Gastroenterology. 1983 Sep;85(3):589-95. PMID 6873605
- [Background] Winston J, Shenoy M, Medley D, Naniwadekar A, Pasricha PJ. The vanilloid receptor initiates and maintains colonic hypersensitivity induced by neonatal colon irritation in rats. Gastroenterology. 2007 Feb;132(2):615-27. doi: 10.1053/j.gastro.2006.11.014. Epub 2006 Nov 10. PMID 17258716
- [Background] Le Gall G, Noor SO, Ridgway K, Scovell L, Jamieson C, Johnson IT, Colquhoun IJ, Kemsley EK, Narbad A. Metabolomics of fecal extracts detects altered metabolic activity of gut microbiota in ulcerative colitis and irritable bowel syndrome. J Proteome Res. 2011 Sep 2;10(9):4208-18. doi: 10.1021/pr2003598. Epub 2011 Aug 8. PMID 21761941
- [Background] Ridlon JM, Kang DJ, Hylemon PB. Bile salt biotransformations by human intestinal bacteria. J Lipid Res. 2006 Feb;47(2):241-59. doi: 10.1194/jlr.R500013-JLR200. Epub 2005 Nov 18. PMID 16299351
- [Background] Wingate DL, Phillips SF, Hofmann AF. Effect of glycine-conjugated bile acids with and without lecithin on water and glucose absorption in perfused human jejunum. J Clin Invest. 1973 May;52(5):1230-6. doi: 10.1172/JCI107290. PMID 4700493
- [Background] De Smet I, Van Hoorde L, Vande Woestyne M, Christiaens H, Verstraete W. Significance of bile salt hydrolytic activities of lactobacilli. J Appl Bacteriol. 1995 Sep;79(3):292-301. doi: 10.1111/j.1365-2672.1995.tb03140.x. PMID 7592123
- [Background] Dussurget O, Cabanes D, Dehoux P, Lecuit M, Buchrieser C, Glaser P, Cossart P; European Listeria Genome Consortium. Listeria monocytogenes bile salt hydrolase is a PrfA-regulated virulence factor involved in the intestinal and hepatic phases of listeriosis. Mol Microbiol. 2002 Aug;45(4):1095-106. doi: 10.1046/j.1365-2958.2002.03080.x. PMID 12180927
- [Background] Stellwag EJ, Hylemon PB. Characterization of 7-alpha-dehydroxylase in Clostridium leptum. Am J Clin Nutr. 1978 Oct;31(10 Suppl):S243-S247. doi: 10.1093/ajcn/31.10.S243. PMID 707382
- [Background] Wells JE, Berr F, Thomas LA, Dowling RH, Hylemon PB. Isolation and characterization of cholic acid 7alpha-dehydroxylating fecal bacteria from cholesterol gallstone patients. J Hepatol. 2000 Jan;32(1):4-10. doi: 10.1016/s0168-8278(00)80183-x. PMID 10673060
- [Background] Wells JE, Williams KB, Whitehead TR, Heuman DM, Hylemon PB. Development and application of a polymerase chain reaction assay for the detection and enumeration of bile acid 7alpha-dehydroxylating bacteria in human feces. Clin Chim Acta. 2003 May;331(1-2):127-34. doi: 10.1016/s0009-8981(03)00115-3. PMID 12691873
- [Background] Kitahara M, Takamine F, Imamura T, Benno Y. Clostridium hiranonis sp. nov., a human intestinal bacterium with bile acid 7alpha-dehydroxylating activity. Int J Syst Evol Microbiol. 2001 Jan;51(Pt 1):39-44. doi: 10.1099/00207713-51-1-39. PMID 11211270
- [Background] Fujita K, Kaku M, Yanagase Y, Ezaki T, Furuse K, Ozawa A, Saidi SM, Sang WK, Waiyaki PG. Physicochemical characteristics and flora of diarrhoeal and recovery faeces in children with acute gastro-enteritis in Kenya. Ann Trop Paediatr. 1990;10(4):339-45. doi: 10.1080/02724936.1990.11747455. PMID 1708960
- [Background] Balamurugan R, Janardhan HP, George S, Raghava MV, Muliyil J, Ramakrishna BS. Molecular studies of fecal anaerobic commensal bacteria in acute diarrhea in children. J Pediatr Gastroenterol Nutr. 2008 May;46(5):514-9. doi: 10.1097/MPG.0b013e31815ce599. PMID 18493205
- [Background] Albert MJ, Bhat P, Rajan D, Maiya PP, Pereira SM, Baker SJ. Faecal flora of South Indian infants and young children in health and with acute gastroenteritis. J Med Microbiol. 1978 May;11(2):137-43. doi: 10.1099/00222615-11-2-137. PMID 660639
- [Background] Boets E, Deroover L, Houben E, Vermeulen K, Gomand SV, Delcour JA, Verbeke K. Quantification of in Vivo Colonic Short Chain Fatty Acid Production from Inulin. Nutrients. 2015 Oct 28;7(11):8916-29. doi: 10.3390/nu7115440. PMID 26516911
- [Background] Camilleri M, Shin A, Busciglio I, Carlson P, Acosta A, Bharucha AE, Burton D, Lamsam J, Lueke A, Donato LJ, Zinsmeister AR. Validating biomarkers of treatable mechanisms in irritable bowel syndrome. Neurogastroenterol Motil. 2014 Dec;26(12):1677-85. doi: 10.1111/nmo.12421. Epub 2014 Sep 22. PMID 25244349
- [Background] Palsson OS, Whitehead WE, van Tilburg MA, Chang L, Chey W, Crowell MD, Keefer L, Lembo AJ, Parkman HP, Rao SS, Sperber A, Spiegel B, Tack J, Vanner S, Walker LS, Whorwell P, Yang Y. Rome IV Diagnostic Questionnaires and Tables for Investigators and Clinicians. Gastroenterology. 2016 Feb 13:S0016-5085(16)00180-3. doi: 10.1053/j.gastro.2016.02.014. Online ahead of print. PMID 27144634
- [Background] Lane DJ, Pace B, Olsen GJ, Stahl DA, Sogin ML, Pace NR. Rapid determination of 16S ribosomal RNA sequences for phylogenetic analyses. Proc Natl Acad Sci U S A. 1985 Oct;82(20):6955-9. doi: 10.1073/pnas.82.20.6955. PMID 2413450
- [Background] Satinsky BM, Gifford SM, Crump BC, Moran MA. Use of internal standards for quantitative metatranscriptome and metagenome analysis. Methods Enzymol. 2013;531:237-50. doi: 10.1016/B978-0-12-407863-5.00012-5. PMID 24060124
- [Background] Caporaso JG, Lauber CL, Walters WA, Berg-Lyons D, Huntley J, Fierer N, Owens SM, Betley J, Fraser L, Bauer M, Gormley N, Gilbert JA, Smith G, Knight R. Ultra-high-throughput microbial community analysis on the Illumina HiSeq and MiSeq platforms. ISME J. 2012 Aug;6(8):1621-4. doi: 10.1038/ismej.2012.8. Epub 2012 Mar 8. PMID 22402401
- [Background] Kozich JJ, Westcott SL, Baxter NT, Highlander SK, Schloss PD. Development of a dual-index sequencing strategy and curation pipeline for analyzing amplicon sequence data on the MiSeq Illumina sequencing platform. Appl Environ Microbiol. 2013 Sep;79(17):5112-20. doi: 10.1128/AEM.01043-13. Epub 2013 Jun 21. PMID 23793624
- [Background] Thomas MC, Thomas DK, Selinger LB, Inglis GD. spyder, a new method for in silico design and assessment of 16S rRNA gene primers for molecular microbial ecology. FEMS Microbiol Lett. 2011 Jul;320(2):152-9. doi: 10.1111/j.1574-6968.2011.02302.x. Epub 2011 May 25. PMID 21554380
- [Background] Schloss PD, Westcott SL, Ryabin T, Hall JR, Hartmann M, Hollister EB, Lesniewski RA, Oakley BB, Parks DH, Robinson CJ, Sahl JW, Stres B, Thallinger GG, Van Horn DJ, Weber CF. Introducing mothur: open-source, platform-independent, community-supported software for describing and comparing microbial communities. Appl Environ Microbiol. 2009 Dec;75(23):7537-41. doi: 10.1128/AEM.01541-09. Epub 2009 Oct 2. PMID 19801464
- [Background] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Background] Gao X, Lin H, Revanna K, Dong Q. A Bayesian taxonomic classification method for 16S rRNA gene sequences with improved species-level accuracy. BMC Bioinformatics. 2017 May 10;18(1):247. doi: 10.1186/s12859-017-1670-4. PMID 28486927
- [Background] McMurdie PJ, Holmes S. Phyloseq: a bioconductor package for handling and analysis of high-throughput phylogenetic sequence data. Pac Symp Biocomput. 2012:235-46. PMID 22174279
- [Background] Tagliacozzi D, Mozzi AF, Casetta B, Bertucci P, Bernardini S, Di Ilio C, Urbani A, Federici G. Quantitative analysis of bile acids in human plasma by liquid chromatography-electrospray tandem mass spectrometry: a simple and rapid one-step method. Clin Chem Lab Med. 2003 Dec;41(12):1633-41. doi: 10.1515/CCLM.2003.247. PMID 14708888
- [Background] Vijayvargiya P, Camilleri M, Shin A, Saenger A. Methods for diagnosis of bile acid malabsorption in clinical practice. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1232-9. doi: 10.1016/j.cgh.2013.04.029. Epub 2013 May 2. PMID 23644387
- [Background] Park J, Kim M, Kang SG, Jannasch AH, Cooper B, Patterson J, Kim CH. Short-chain fatty acids induce both effector and regulatory T cells by suppression of histone deacetylases and regulation of the mTOR-S6K pathway. Mucosal Immunol. 2015 Jan;8(1):80-93. doi: 10.1038/mi.2014.44. Epub 2014 Jun 11. PMID 24917457
- [Background] Dall'Amico R, Montini G, Pisanello L, Piovesan G, Bottaro S, Cracco AT, Zacchello G, Zacchello F. Determination of inulin in plasma and urine by reversed-phase high-performance liquid chromatography. J Chromatogr B Biomed Appl. 1995 Oct 6;672(1):155-9. doi: 10.1016/0378-4347(95)00209-2. PMID 8590929
- [Background] Heaton KW, Radvan J, Cripps H, Mountford RA, Braddon FE, Hughes AO. Defecation frequency and timing, and stool form in the general population: a prospective study. Gut. 1992 Jun;33(6):818-24. doi: 10.1136/gut.33.6.818. PMID 1624166
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Benjamini Y and Y. Hochberg. Controlling the false discovery rate: a practical and powerful approach to multiple testing. Journal of the Royal Statistical Society 1995. Series B 57:289-300